CLINICAL TRIAL: NCT04497909
Title: The Impact of Online Mindfulness on Depression, Anxiety, Stress and Burnout in Medical Students and Residents
Brief Title: Online Mindfulness for Medical Trainees
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The online mindfulness is no longer being offered and recruitment can no longer happen.
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00103222
Record Dates: First submitted 2020-07-30; First posted 2020-08-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Stress; Anxiety; Depression; Mindfulness
Keywords: Mindfulness; Medical Students; Medical Residents; Medical Trainees
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: The three groups of participants are a pre-clerkship cohort consisting of first- and second-year medical students, a clerkship cohort consisting of third- and fourth-year medical students and the third cohort consisting of medical residents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-clerkship cohort (Experimental): First- and second-year medical students
  Interventions: Behavioral: Mindfulness
- Clerkship cohort (Experimental): Third- and fourth-year medical students
  Interventions: Behavioral: Mindfulness
- Resident cohort (Experimental): Medical residents
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Mindfulness online training

SUMMARY:
Medical students and medical residents are subject to increased stressors throughout their education. There is increased depression, anxiety, burnout, and distress in medical trainees compared to the general population. Globally, roughly 3 out of 10 medical students experience anxiety. A recent study also found that almost 3 out of 10 medical trainees experience depression or depressive symptoms and approximately 1 out of 10 have suicidal thoughts. All of this leads to poorer academics, increased dropout rates as well as reduced empathy and quality of care in affected trainees.

Mindfulness programs are increasingly being used in medical schools to help deal with increased levels of depression, anxiety, stress, and burnout. Several studies have looked at medical students, medical residents, and various other healthcare professionals. These programs have been found to reduce depression, anxiety and stress while significantly improving mood, well being and mindfulness.

Although in-person mindfulness programs have shown several benefits, there are limitations to its use in medical programs. A lack of time, flexibility, accessibility as well as the issue of cost, impact the uptake of in-person mindfulness programs. A potential alternative to this is online mindfulness programs. To date, there is limited research regarding medical students and online mindfulness programs. With that being said, studies focussed on other populations and online mindfulness have shown reductions in depression, anxiety and stress with improvements in mindfulness and mood.

The study being proposed involves providing online mindfulness to medical students and residents in an 8-week program that consists of 8, 1-hour sessions with a mindfulness coach. Participants will be enrolled through informed consent. All participants will be given pre and post participation questionnaires to examine the impact of online mindfulness on anxiety, depression, stress and burnout. The results of this research may lead to future studies looking at the impact of online mindfulness practice for medical trainees and might also help open up the possibility of offering such programs in medical schools.

DETAILED DESCRIPTION:
BACKGROUND

The transition to medical school and the subsequent years that follow are a period of increased stress on trainees. Research shows that there is a higher prevalence of depression, anxiety and burnout amongst U.S. and Canadian medical students compared to the general population. In addition, distress is consistently higher in medical trainees compared to the general population and in age matched non-medical students. A recent systematic review found the prevalence of depression or depressive symptoms in medical trainees to be 27.2% and suicidal ideation to be 11.1%. A separate systematic review found that the prevalence of anxiety in medical students was 33.8% globally. Increased levels of distress and anxiety lead to poorer academics and increased dropout rates, as well as a reduced empathy, enthusiasm, and quality of care.

An intervention that has been gaining traction in recent years to manage the psychological strain placed on medical trainees is mindfulness training. A study of 140 second year medical students participating in a 10-week mindfulness-based stress reduction program reported significant improvement in mood and reduced psychological distress. Similar results have been found in randomised controlled trials with health care professionals as well as surgical and psychiatric residents. Furthermore, a 2017 systematic review of 19 papers looking at the effectiveness of mindfulness interventions in healthcare professionals found them to decrease stress, anxiety and depression while improving mindfulness, empathy and mood. These benefits may potentially continue over the long term based on results from a 2018 longitudinal study of mindfulness training in medical and psychology students. At the six year follow up with the intervention group, they reported increased well being, mindfulness, and problem-focused coping.

Although in-person mindfulness training has shown several benefits, there are limitations to implementing these programs in the demanding schedules of medical trainees. In addition to a lack of time, flexibility, costs, anonymity, and accessibility may limit its effectiveness as well. A modality that may reduce these limitations is online mindfulness. This format allows flexibility with regards to when trainees would be able to access the material, it would be more cost effective and could be accessed from rural and remote areas as suggested in a 2020 pilot study completed with Australian rural medical students. Results indicated significant reduction in perceived stress and increases in self compassion 4 months after the 8-week online mindfulness program. Online mindfulness interventions have been studied in several other populations and a 2016 meta analysis of 15 randomised controlled trials, found online mindfulness interventions to reduce depression, anxiety, and stress with an associated increase in well being and mindfulness.

To date, there is limited research looking at online mindfulness as a tool for medical students and residents. The study being proposed here, would assess the impact of an online mindfulness intervention on medical trainees with regards to depression, anxiety, stress, burnout, and mindfulness.

OBJECTIVE

To explore the potential benefits of online mindfulness on depression, anxiety, stress, and burnout in medical trainees.

To explore the changes in mindfulness level over the course of an online mindfulness program offered to medical trainees.

HYPOTHESIS

The investigators hypothesize that medical students and residents that participate in the online mindfulness program will report reduced depression, stress, anxiety, and burnout as well as improved mindfulness.

MATERIALS AND METHODS

This study is a prospective observational study.

Procedure

Following recruitment, all participants will complete a general demographic form as well as four scales that measure depression, anxiety, stress, burnout, and mindfulness. The same four scales will be completed by all participants at the end of the mindfulness training and 3 months after the training.

Online Mindfulness Intervention (OMI)

All participants will be instructed by a mindfulness practitioner/coach online through 8, 1-hour sessions over the course of eight weeks. Trainees will have the ability to retrieve the online sessions at their convenience. Weekly journals will be provided to measure attendance and frequency and duration of mindfulness practice.

Instruments

General Demographic Form: A researcher created demographic data form (age, educational level, prior experience with mindfulness, history of depression and anxiety) to be completed by the medical trainees at enrolment.

Depression, Anxiety and Stress Scale: 21 item Depression, Anxiety, Stress Scale to be completed by the medical trainees at three time points.

Oldenburg Burnout Inventory for Students: 16 item scale to measure burnout in students completed at three time points.

Mindfulness Scales: 15 item Mindfulness Attention Awareness Scale and the 13 item Toronto Mindfulness Scale will be completed by the medical trainees at three time points.

Mindfulness Weekly Journal: Document recording the duration and frequency of mindfulness practice during the study to assess attendance to the online class.

DATA ANALYSIS

Study data will be managed using Research Electronic Data Capture, a secure, web-based software platform, hosted at the University of Alberta. Group demographics will be compared with t-test, chi-square and Mann-Whitney U as appropriate. The scores of the four questionnaires will be analyzed with the Wilcoxon Signed-Rank test for within group comparison. The Spearman correlation test will be used for correlation between the mindfulness scores and the stress, anxiety, depression, and burnout scores. 2-tailed p-values will be used.

ELIGIBILITY:
Inclusion Criteria:

- A medical trainee who registered for the online mindfulness elective

Exclusion Criteria:

- None

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Change in stress symptoms time 1 | Change from recruitment to immediately after the online mindfulness course
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of stress symptoms. Minimum score is 0. Maximum score is 21.
Change in stress symptoms time 2 | Change from recruitment to 3 months after the online mindfulness course
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of stress symptoms. Minimum score is 0. Maximum score is 21.
Change in anxiety symptoms time 1 | Change from recruitment to immediately after the online mindfulness course
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of anxiety symptoms. Minimum score is 0. Maximum score is 21.
Change in anxiety symptoms time 2 | Change from recruitment to 3 months after the online mindfulness course
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of anxiety symptoms. Minimum score is 0. Maximum score is 21.
Change in depression symptoms time 1 | Change from recruitment to immediately after the online mindfulness course
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of depression symptoms. Minimum score is 0. Maximum score is 21.
Change in depression symptoms time 2 | Change from recruitment to 3 months after the online mindfulness course
  using the Depression Anxiety Stress Scale -21. Scores for individual question range from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). A high score means a higher level of depression symptoms. Minimum score is 0. Maximum score is 21.
Change in burnout symptoms time 1 | Change from recruitment to immediately after the online mindfulness course
  using the Oldenburg Burnout Inventory for Students; a 16 item scale to measure burnout. Scores for individual question range from 1 (strongly disagree) to 4 (strongly agree). A high score means a higher level of burnout symptoms. This scale has 2 subscales. Minimum score is 8. Maximum score is 32 for both subscales.
Change in burnout symptoms time 2 | Change from recruitment to 3 months after the online mindfulness course
  using the Oldenburg Burnout Inventory for Students; a 16 item scale to measure burnout. Scores for individual question range from 1 (strongly disagree) to 4 (strongly agree). A high score means a higher level of burnout symptoms. This scale has 2 subscales. Minimum score is 8. Maximum score is 32 for both subscales.
Change in mindful awareness time 1 | Change from recruitment to immediately after the online mindfulness course
  using the Mindfulness Attention Awareness Scale. Scores for individual question range from 1 (Almost Never) to 6 (Almost Always). Minimum score is 15. Maximum score is 90.
  And using Toronto Mindfulness Scale. Scores for individual question range from 0 (Not at all) to 4 (Very much). This scale has 2 subscales. Minimum score is 0. Maximum score is 24 for the first subscale and 28 for the second subscale.
  A high score in both scales (and subscales)means a high mindful awareness level.
Change in mindful awareness time 2 | Change from recruitment to 3 months after the online mindfulness course
  using the Mindfulness Attention Awareness Scale. Scores for individual question range from 1 (Almost Never) to 6 (Almost Always). Minimum score is 15. Maximum score is 90.
  And using Toronto Mindfulness Scale. Scores for individual question range from 0 (Not at all) to 4 (Very much). This scale has 2 subscales. Minimum score is 0. Maximum score is 24 for the first subscale and 28 for the second subscale.
  A high score in both scales (and subscales)means a high mindful awareness level.

SECONDARY OUTCOMES:
Frequency of Mindfulness practice 1 | From recruitment to the end of the online mindfulness elective (8 weeks in total)
  Frequency of mindfulness practice
Duration of Mindfulness practice 1 | From recruitment to the end of the online mindfulness elective (8 weeks in total)
  Duration of mindfulness practice
Frequency of Mindfulness practice 2 | From the end of the online mindfulness elective until three months after
  Frequency of mindfulness practice
Duration of Mindfulness practice 2 | From the end of the online mindfulness elective until three months after
  Duration of mindfulness practice

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine Landry, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No